CLINICAL TRIAL: NCT07106515
Title: Development of Taxi Teaching for Strangled Inguinal Hernias in Children
Acronym: DETHREAT
Status: Not yet recruiting | Type: Observational
Sponsor: University Hospital, Angers (Other Government)
Responsible Party: Sponsor
Other Study IDs: 49RC25_0085
Record Dates: First submitted 2025-07-30; First posted 2025-08-06 (Actual); Last update posted 2025-08-06 (Actual); Status verified 2025-07

CONDITIONS: Pediatric Inguinal Hernia
Keywords: Strangulated hernia; External hernia reduction maneuver

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- patients before doctors were trained in hernia reduction procedures
- patients after doctors were trained in hernia reduction procedures

SUMMARY:
Inguinal hernias in children are very common but pose a risk of strangulation, which, if not treated quickly, can lead to life-threatening complications (intestinal obstruction, peritonitis) or functional complications (testicular ischemia). The manual reduction of a strangulated inguinal hernia, known as taxis, is often unfamiliar to the first doctors to see the child, whether they are general practitioners, pediatricians, or emergency physicians, and therefore requires second- or third-line treatment, which prolongs the delay in care and increases the risk of serious complications. The hypothesis is that targeted professional training using mannequins to practice this reduction maneuver for the doctors concerned would reduce the time required for reduction and thus improve the care of these patients. To this end, and in the absence of a dedicated model on the market for medical education through simulation, investigatores are developing a pediatric manikin to train doctors in performing hernia reduction maneuvers.

The aim of this study is therefore to compare the care pathway for children with strangulated inguinal hernias before and after training on mannequins for doctors in therapeutic taxis, in order to demonstrate in real life the impact of procedural training through simulation on improving patient care.

DETAILED DESCRIPTION:
The objective is to show that a better understanding of hernia reduction techniques by frontline physicians leads to a reduction in the time taken to reduce strangulated inguinal hernias in children consulting for this reason. Investigators will therefore compare the time taken to reduce the hernia before and after the doctors concerned learned the reduction procedure, in the population of children treated for strangulated inguinal hernias in a pediatric surgery department of the HUGO network (Hôpitaux Universitaire du Grand Ouest - University Hospitals of western France). The study will therefore be divided into two phases: an initial retrospective, multicenter phase covering the period prior to the training of physicians in hernia reduction techniques, followed by a prospective, multicenter phase covering the period after training.

ELIGIBILITY:
Inclusion Criteria:

* Any child (pediatric population defined as under 16 years of age) presenting at a university hospital or hospital in western France with a clinical diagnosis of strangulated inguinal hernia

Exclusion Criteria:

* Refusal to participate in the search for legal representatives
* Differential diagnosis of strangulated inguinal hernia (adenopathy, cord cyst, cryptorchid testicle, unstrangulated hernia)
* Patients and/or parents who do not speak French
* Patients not affiliated with a social security system.

Max Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Children with strangulated inguinal hernia presenting at hospital in western France
Sampling Method: Non-Probability Sample
Enrollment: 104 (Estimated)
Dates: Start 2025-11-01 (Estimated); Primary Completion 2029-11-01 (Estimated); Study Completion 2030-04-01 (Estimated)

PRIMARY OUTCOMES:
Hernia reduction time | 6 month
  hernia reduction time in children with stranglutated hernia presenting in a hospital of western France before and after the doctors learned the reduction hernia maneuver.

SECONDARY OUTCOMES:
Overal success rate of hernia reduction | 6 month
  The overall success rate of hernia reduction by external reduction maneuver based on the status of the operator (having participated in training or not having participated in training)

CONTACTS AND LOCATIONS:
Overall Officials: Louise RENOULT, Study Chair — University Hospital of Angers

IPD SHARING:
Plan to Share IPD: Undecided